CLINICAL TRIAL: NCT03001687
Title: Impact of Vitamin D Enteral Supplementation on Hepcidin Serum Levels and Transfusion Requirements in Surgical and Critically Ill Patients
Brief Title: Impact of Vitamin D Supplementation on Hepcidin Levels and Transfusion Requirements in Surgical and Septic Patients
Acronym: DEHEPTRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Cristina Petrisor, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 434/24.11.2016
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis; Surgical Injuries
Keywords: hepcidin; sepsis; surgery; vitamin D
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Intraoperative Complications | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D + (Experimental): Patients in the "vitamin D" group will receive enteral supplementation with vitamin D, blood collection 3mL is performed in the first 24 hours after admission and one week later for serum hepcidin measurement
  Interventions: Dietary Supplement: enteral supplementation with vitamin D; Other: blood collection 3mL
- vitamin D - (Placebo Comparator): Patients in "vitamin D -" group do not receive enteral supplementation with vitamin D and represent the control group, blood collection 3mL is performed in the first 24 hours after admission and one week later for serum hepcidin measurement
  Interventions: Other: blood collection 3mL

INTERVENTIONS:
Dietary Supplement: enteral supplementation with vitamin D — Patients allocated to the "vitamin D +" group receive enteral supplementation with high-dose vitamin D (250.000UI)
  Arms: vitamin D +
Other: blood collection 3mL — all patients will have hepcidin levels measured in the first 24 hours after admission and one week after

SUMMARY:
Acute inflammation induced by surgery and sepsis is complicated by the development of iron-restricted anemia due to the up-regulation of hepcidin. Excess hepcidin causes intracellular sequestration of iron, decreasing its availability for erythropoiesis. Hepcidin might be a potential target to reduce transfusion requirements in surgical and sepsis patients. Vitamin D supplementation might constitute a novel strategy to modulate the hepcidin-ferroportin-iron axis. Up to now, there are no data regarding the possibility that by using vitamin D supplementation in surgical and septic shock patients, the physicians could ameliorate anemia and, hence, reduce transfusion requirements. Aim: to conduct a randomised controlled trial to determine the impact of high-dose vitamin D enteral supplementation on serum hepcidin levels and transfusion requirements after major abdominal surgery and in septic shock patients.

DETAILED DESCRIPTION:
Patient blood management has become an important concept for the perioperative care of the surgical patients and in septic patients, aiming to improve outcomes. Hepcidin might be a potential target to reduce transfusion requirements after major abdominal surgery and in patients with sepsis. Major surgery and sepsis induce complex immune dysregulations, characterised by a pro-inflammatory state (the postoperative acute-phase reaction). Excess hepcidin values in acute inflammatory conditions might represent an exaggerated response that leads to iron-sequestration anemia, a functional iron deficiency anemia. Vitamin D supplementation might constitute a novel strategy to modulate the hepcidin-ferroportin-iron axis in surgery and sepsis-induced acute inflammation. Thus, vitamin D might impact hepcidin values and might reduce transfusion requirements.

I. Inflammation-induced regulation of the hepcidin-ferroportin-iron axis

Surgery and sepsis are associated with iron-restricted anemia. After major abdominal surgery and sepsis, a prototypical inflammatory syndrome, often complicated by the development of anemia, appears. Inflammatory cytokines (like interleukin 6) released during acute infection alter iron metabolism by inducing excess synthesis of hepcidin. Anemia after major abdominal surgery and sepsis may be the expression of impaired erythropoiesis as a result of hepcidin up-regulation. Hepcidin plays a role in the development of anemia, together with the inhibition of erythropoietin production, a decreased lifespan of erythrocytes, and a blunted erythropoietic response. Functional iron deficiency is increasingly recognised as a cause of anemia in the general surgical patient and in patients with sepsis.

Iron is a two-faced element. First, iron is essential for living as it is incorporated in the "breathing" molecule haemoglobin and in the mitochondrial respiratory chain. On the other hand, iron is detrimental due to the generation of oxidative stress and its availability for the growing of bacteria. Low serum iron level is considered detrimental as it leads to anemia and low tissue oxygen delivery. Iron deficiency and anemia are associated with poor outcomes in surgical and septic patients. Also, transfusion is associated with immune suppression and other adverse reactions. Thus, other approaches to the correction of anemia are advocated, even though not yet included in the clinical practice.

Hepcidin is the master regulator of iron metabolism and hence, a modulator of anemia in states of inflammation. Hepcidin is an acute phase protein synthetised in the liver and which acts as an hyposideremia inducing hormone. It binds to ferroportin (an iron exporter) and prevents the release of iron from the cells: prevents the absorption of dietary iron from enterocytes and prevents iron release from macrophages, where it is stored. Thus, the effect of hepcidin would be iron sequestration, lowering the serum iron concentrations. The beneficial result would be a low availability of iron for bacterial growth (thus, a direct antimicrobial effect) and less oxidative stress. The detrimental result is the limited possibility for the synthesis of new haemoglobin molecules and the occurrence of anemia. The up-regulation of hepcidin, as a pro-inflammatory biomarker, characterises both acute and chronic inflammatory conditions. The induction of hepcidin synthesis may be the cause for the iron-restricted erythropoiesis in the surgical population and in patients with sepsis. The induction of hepcidin synthesis may contribute to the development of anemia, which is detrimental for tissue oxygenation and might increase transfusion requirements and the aggravation of immune suppression after blood transfusion. In animal models of anemia due to inflammation, hepcidin knockout mice had milder anemia and faster recovery.

Excess values of the iron regulating hormone hepcidin causes intracellular sequestration of iron and might decrease the availability of iron for erythropoiesis, leading to the anemia frequently encountered in inflammatory conditions. Anemia is not only very frequent among critically ill patients, but is associated with increased transfusion rates and worse outcomes. Anemia may impair oxygen delivery to peripheral tissues and impose transfusion, which itself carries the risk of further immune suppression. Recent data has emphasised the need to restrict transfusions as much as possible, as transfusion is associated with increased morbidity and mortality. Instead, alternative methods to improve anemia and ameliorate tissue oxygen delivery might be beneficial.

II. Vitamin D down-regulates hepcidin expression

Vitamin D is a hormone promoting bone health, which also has a wide range of cellular activities including the differentiation of hematopoietic cells and down-regulation of inflammatory cytokines. Vitamin D has anti-inflammatory and immune-regulating properties and the maintenance of adequate vitamin D status may play a role in managing inflammation and immunity. Vitamin D supplementation in patients with chronic inflammatory conditions like chronic kidney disease improves the values of circulating markers of inflammation and immunity. Recently, it has been highlighted that in certain conditions, like chronic kidney disease, the administration of vitamin D reduces serum hepcidin values and transfusion requirements.

Up to now, there are no data regarding the possibility that by using vitamin D supplementation in surgical or septic shock patients, the physicians could target the hepcidin-ferroportin-iron axis to prevent the occurrence of anemia and, hence, reduce transfusion requirements. Oral vitamin D supplementation lowers hepcidin values and might increase erythropoiesis and decrease inflammation.

III. Vitamin D supplementation in the critically ill. Safety profile

The therapeutic potential of vitamin D is a topic of intense interest. A high prevalence of low vitamin D levels has been confirmed in patients who are critically ill. Vitamin D deficiency is associated with higher infection rates, 30-day mortality and in-hospital mortality in adult critically ill patients. During critical illness, vitamin D supplementation has a favorable safety profile and a possible mechanism of vitamin D supplementation in inducing bactericidal pleiotropic effects has been suggested. To improve vitamin D status, high-dose vitamin D is required in the critically ill, as they display a blunted response to supplementation. Recent evidence suggests that treatment of vitamin-D deficient critically ill patients may improve outcomes and mortality, possibly through enhancing innate immunity and the inhibition of proinflammatory cytokines. Further clinical trials to explore the effects of vitamin D supplementation on the up-regulation process of proinflammatory cytokines are needed.

ELIGIBILITY:
Inclusion Criteria:

* sepsis and septic shock patients
* patients with major abdominal surgery

Exclusion Criteria:

* chronic inflammatory conditions (chronic kidney disease, hematologic, and rheumatic/autoimmune disease)
* morbid obesity (BMI over 40kg/m2)
* pregnancy and lactation
* hypercalcemia (total calcium> 10.6mg/dL, serum ionized calcium>5.4mg/dL)
* tuberculosis, sarcoidosis
* nephrolithiasis
* recent history of vitamin D supplementation or erythropoietin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hepcidin concentration (ng/mL) | one week after intervention
  Hepcidin serum concentrations measured one week after the intervention

SECONDARY OUTCOMES:
Number of Packed red cells | two weeks after intervention
  The number of transfused packed red cells in the first two weeks after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Petrisor, MD, PhD, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu Cluj-Napoca
Locations (1):
- Iuliu Hatieganu University of Medicine and Pharmacy Cluj-Napoca, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No
Only on request

REFERENCES:
- [Background] Lasocki S, Longrois D, Montravers P, Beaumont C. Hepcidin and anemia of the critically ill patient: bench to bedside. Anesthesiology. 2011 Mar;114(3):688-94. doi: 10.1097/ALN.0b013e3182065c57. No abstract available. PMID 21258235
- [Background] Clevenger B, Richards T. Pre-operative anaemia. Anaesthesia. 2015 Jan;70 Suppl 1:20-8, e6-8. doi: 10.1111/anae.12918. PMID 25440391
- [Background] Heming N, Montravers P, Lasocki S. Iron deficiency in critically ill patients: highlighting the role of hepcidin. Crit Care. 2011;15(2):210. doi: 10.1186/cc9992. Epub 2011 Mar 22. No abstract available. PMID 21457511
- [Background] Lasocki S, Gaillard T, Rineau E. Iron is essential for living! Crit Care. 2014 Dec 8;18(6):678. doi: 10.1186/s13054-014-0678-7. PMID 25673336
- [Background] Heming N, Letteron P, Driss F, Millot S, El Benna J, Tourret J, Denamur E, Montravers P, Beaumont C, Lasocki S. Efficacy and toxicity of intravenous iron in a mouse model of critical care anemia*. Crit Care Med. 2012 Jul;40(7):2141-8. doi: 10.1097/CCM.0b013e31824e6713. PMID 22564959
- [Background] Zeng C, Chen Q, Zhang K, Chen Q, Song S, Fang X. Hepatic hepcidin protects against polymicrobial sepsis in mice by regulating host iron status. Anesthesiology. 2015 Feb;122(2):374-86. doi: 10.1097/ALN.0000000000000466. PMID 25264597
- [Background] Kali A, Charles MV, Seetharam RS. Hepcidin - A novel biomarker with changing trends. Pharmacogn Rev. 2015 Jan-Jun;9(17):35-40. doi: 10.4103/0973-7847.156333. PMID 26009691
- [Background] Ruchala P, Nemeth E. The pathophysiology and pharmacology of hepcidin. Trends Pharmacol Sci. 2014 Mar;35(3):155-61. doi: 10.1016/j.tips.2014.01.004. Epub 2014 Feb 17. PMID 24552640
- [Background] Kim A, Fung E, Parikh SG, Valore EV, Gabayan V, Nemeth E, Ganz T. A mouse model of anemia of inflammation: complex pathogenesis with partial dependence on hepcidin. Blood. 2014 Feb 20;123(8):1129-36. doi: 10.1182/blood-2013-08-521419. Epub 2013 Dec 19. PMID 24357728
- [Background] Meybohm P, Shander A, Zacharowski K. Should we restrict erythrocyte transfusion in early goal directed protocols? BMC Anesthesiol. 2015 May 9;15:75. doi: 10.1186/s12871-015-0054-4. PMID 25956725
- [Background] Shah A, Stanworth SJ, McKechnie S. Evidence and triggers for the transfusion of blood and blood products. Anaesthesia. 2015 Jan;70 Suppl 1:10-9, e3-5. doi: 10.1111/anae.12893. PMID 25440390
- [Background] Sadaka F, Trottier S, Tannehill D, Donnelly PL, Griffin MT, Bunaye Z, O'Brien J, Korobey M, Lakshmanan R. Transfusion of red blood cells is associated with improved central venous oxygen saturation but not mortality in septic shock patients. J Clin Med Res. 2014 Dec;6(6):422-8. doi: 10.14740/jocmr1843w. Epub 2014 Sep 9. PMID 25247015
- [Background] Sun CC, Vaja V, Chen S, Theurl I, Stepanek A, Brown DE, Cappellini MD, Weiss G, Hong CC, Lin HY, Babitt JL. A hepcidin lowering agent mobilizes iron for incorporation into red blood cells in an adenine-induced kidney disease model of anemia in rats. Nephrol Dial Transplant. 2013 Jul;28(7):1733-43. doi: 10.1093/ndt/gfs584. Epub 2013 Jan 22. PMID 23345622
- [Background] Alvarez JA, Zughaier SM, Law J, Hao L, Wasse H, Ziegler TR, Tangpricha V. Effects of high-dose cholecalciferol on serum markers of inflammation and immunity in patients with early chronic kidney disease. Eur J Clin Nutr. 2013 Mar;67(3):264-9. doi: 10.1038/ejcn.2012.217. Epub 2013 Jan 30. PMID 23361158
- [Background] Smith EM, Tangpricha V. Vitamin D and anemia: insights into an emerging association. Curr Opin Endocrinol Diabetes Obes. 2015 Dec;22(6):432-8. doi: 10.1097/MED.0000000000000199. PMID 26414080
- [Background] Zughaier SM, Alvarez JA, Sloan JH, Konrad RJ, Tangpricha V. The role of vitamin D in regulating the iron-hepcidin-ferroportin axis in monocytes. J Clin Transl Endocrinol. 2014 Mar 21;1(1):19-25. doi: 10.1016/j.jcte.2014.01.003. PMID 25097830
- [Background] Bacchetta J, Zaritsky JJ, Sea JL, Chun RF, Lisse TS, Zavala K, Nayak A, Wesseling-Perry K, Westerman M, Hollis BW, Salusky IB, Hewison M. Suppression of iron-regulatory hepcidin by vitamin D. J Am Soc Nephrol. 2014 Mar;25(3):564-72. doi: 10.1681/ASN.2013040355. Epub 2013 Nov 7. PMID 24204002
- [Background] Han JE, Ziegler TR. Vitamin D supplementation in sepsis and critical illness: where are we now? Am J Respir Crit Care Med. 2014 Sep 1;190(5):483-5. doi: 10.1164/rccm.201408-1443ED. No abstract available. PMID 25171307
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] Quraishi SA, Bittner EA, Blum L, McCarthy CM, Bhan I, Camargo CA Jr. Prospective study of vitamin D status at initiation of care in critically ill surgical patients and risk of 90-day mortality. Crit Care Med. 2014 Jun;42(6):1365-71. doi: 10.1097/CCM.0000000000000210. PMID 24557421
- [Background] de Haan K, Groeneveld AB, de Geus HR, Egal M, Struijs A. Vitamin D deficiency as a risk factor for infection, sepsis and mortality in the critically ill: systematic review and meta-analysis. Crit Care. 2014 Dec 5;18(6):660. doi: 10.1186/s13054-014-0660-4. PMID 25475621
- [Background] Upala S, Sanguankeo A, Permpalung N. Significant association between vitamin D deficiency and sepsis: a systematic review and meta-analysis. BMC Anesthesiol. 2015 Jun 4;15:84. doi: 10.1186/s12871-015-0063-3. PMID 26041306
- [Background] Venkatesh B, Nair P. Hypovitaminosis D and morbidity in critical illness: is there proof beyond reasonable doubt? Crit Care. 2014 May 8;18(3):138. doi: 10.1186/cc13863. PMID 24976501
- [Background] Dickerson RN, Berry SC, Ziebarth JD, Swanson JM, Maish GO 3rd, Minard G, Brown RO. Dose-response effect of ergocalciferol therapy on serum 25-hydroxyvitamin D concentration during critical illness. Nutrition. 2015 Oct;31(10):1219-23. doi: 10.1016/j.nut.2015.03.008. Epub 2015 Apr 4. PMID 26213135
- [Background] Nair P, Venkatesh B, Lee P, Kerr S, Hoechter DJ, Dimeski G, Grice J, Myburgh J, Center JR. A Randomized Study of a Single Dose of Intramuscular Cholecalciferol in Critically Ill Adults. Crit Care Med. 2015 Nov;43(11):2313-20. doi: 10.1097/CCM.0000000000001201. PMID 26186566
- [Background] Christopher KB. Vitamin D supplementation in the ICU patient. Curr Opin Clin Nutr Metab Care. 2015 Mar;18(2):187-92. doi: 10.1097/MCO.0000000000000147. PMID 25635597
- [Background] Leaf DE, Raed A, Donnino MW, Ginde AA, Waikar SS. Randomized controlled trial of calcitriol in severe sepsis. Am J Respir Crit Care Med. 2014 Sep 1;190(5):533-41. doi: 10.1164/rccm.201405-0988OC. PMID 25029202
- [Background] Smith EM, Alvarez JA, Kearns MD, Hao L, Sloan JH, Konrad RJ, Ziegler TR, Zughaier SM, Tangpricha V. High-dose vitamin D3 reduces circulating hepcidin concentrations: A pilot, randomized, double-blind, placebo-controlled trial in healthy adults. Clin Nutr. 2017 Aug;36(4):980-985. doi: 10.1016/j.clnu.2016.06.015. Epub 2016 Jun 27. PMID 27402475